CLINICAL TRIAL: NCT02397356
Title: Inhaled Nebulised S(+)-Ketamine for Postoperative Analgesia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of study personnel
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R14066M; 2014-000837-22 (EudraCT Number)
Record Dates: First submitted 2014-12-01; First posted 2015-03-24 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative
Keywords: ketamine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine first AB (Experimental): Patients in this group will first receive a dose of ketamine in the nebulised form when they ask for pain relief. The second time they ask for pain relief, they will receive physiological salt in the nebulised form.
  Interventions: Drug: Ketamine first AB; Drug: Placebo first BA
- Placebo first BA (Active Comparator): Patients in this group will first receive physiological salt in the nebulised form form when they ask for pain relief. The second time they ask for pain relief, they will receive a dose of ketamine in the nebulised.
  Interventions: Drug: Ketamine first AB; Drug: Placebo first BA

INTERVENTIONS:
Drug: Ketamine first AB — Nebulised ketamine 1mg/kg
  Other Names: S(+)-ketamine
Drug: Placebo first BA — Nebulised saline 1-2ml
  Other Names: NaCl; Saline

SUMMARY:
Ketamine has been administrated via the intravenous, intramuscular, subcutaneous, rectal, oral, transdermal, intranasal, sublingual, transmucosal, epidural, intrathecal, and intra-articular routes. Pharmacokinetic properties of inhaled ketamine have not been studied officially, but one of the investigators researchers has tested nebulized ketamine on himself with repeated painful stimulus and monitoring applied. Based on this experiment, analgesic effect is roughly estimated to begin in 3 minutes.Ketamine has been used successfully to treat acute pain in intranasal form. The primary purpose of this study is to evaluate whether nebulised S(+)-ketamine carries potential as a an analgesic bypassing first pass metabolism and without the need for intravenous access. Secondary aim is to assess the duration of analgesia obtained by nebulized S-ketamine. Thirdly, the aim is to evaluate whether inhaled nebulized ketamine decreases the need for rescue analgesia during PACU care. The subjects are recruited among patients coming in for a surgical intervention (orthopedic, gastrointestinal, plastic or urologic surgery) and needing further observation in postoperative care unit (PACU).

It was calculated that sample size of 8 subjects per group would be required to achieve statistical power of 80% and detect a difference of 3 units in NRS-values with standard deviation of 2 units and type I error of 5%. To prepare for possible dropouts, total of 20 subjects will be recruited (10 in each group).

Patients will receive either nebulized placebo (i.e. saline) or ketamine (Ketanest-S) when they require pain alleviation in the PACU. Dosage of ketamine is 1 mg/kg. Patients will be randomized into two groups so that other group's first inhalation contains ketamine and second inhalation placebo and in the opposite order.

DETAILED DESCRIPTION:
Introduction

Since first described in 1965 1, the phencyclidine derivative ketamine [(RS)-2-(2-Chlorophenyl)-2-(methylamino)cyclohexanone] has gained widespread use as an anaesthetic, sedative and analgesic. 2 There is some evidence that ketamine might possess antidepressant effects as well. 3 In anaesthetic dosages, ketamine produces dissociative anaesthesia with low respiratory or circulatory depressive effects. Therefore it is the optimal anaesthetic e.g. in haemodynamically compromised patients or when minimal respiratory depression is desirable during induction of anaesthesia, e.g. in emergency care. 2 Despite this, adverse psychomimetic effects such as hallucinations and initially observed effects on intracranial pressure (ICP) have limited the use of ketamine without additional sedation or in patients with neurological injury. 4 Increasing evidence, however, supports the notion that - during controlled ventilation - ketamine can be safely used in patients with neurotrauma 5 and that the adverse psychometric side effects are less pronounced with the S(+)-enantiomer. 6,7

Both chiral forms of ketamine modulate nociception mainly via inhibition of N-methyl-D-aspartate (NMDA)-receptor activation. 8 Analgesic effect is also related to modulation of signalling via nitric oxide (NO) synthase inhibition 4,9, monoamine 10,11 and muscarinic 12 neurotransmission, and µ-, δ- and κ-opiate receptor agonism 13.

S(+)-ketamine has been observed to exert analgesic effect two-to-four times that of racemic ketamine 17 or the R(-)-isomer 18 alone. Although observations regarding unwanted psychometric effects with equianalgetic dosages of the S(+)-enantiomer and racemic ketamine are in favour of S(+)-ketamine 6,7 or controversial 17,18, it would seem that the superior potency 17 and shorter duration of effect 19 of the S(+)-ketamine allows for easier dosing and titration.

Ketamine has been administrated via the intravenous, intramuscular, subcutaneous, rectal, oral, transdermal, intranasal, sublingual, transmucosal, epidural, intrathecal, and intra-articular routes. 20-30 Following intravenous administration, bioavailability is 90 % and peak anaesthetic effect is observed in 1 to 5 minutes. 2 Parenteral administration results in more effective analgesia due to avoidance of first-pass metabolism in the liver to the less potent norketamine, but, on the other hand, oral administration may result in less psychometric side effects as norketamine does not exert hallucinogenic properties. 2 Pharmacokinetic properties of inhaled ketamine have not been studied officially, but one of our researchers has tested nebulized ketamine on himself with repeated painful stimulus and monitoring applied. Based on this experiment, analgesic effect is roughly estimated to begin in 3 minutes.

Ketamine is metabolised in the liver via cytochrome (CYP2B6, CYP3A4 and CYP2C9) -enzyme pathways. 14,15 An active metabolite of ketamine - norketamine - possesses the potency of approximately one-third that of ketamine. Ketamine metabolites are renally excreted with an elimination half-life of approximately 2-3 hours. 16

Ketamine has been used successfully to treat acute pain in intranasal form. Studies in prehospital and emergency department settings have concluded that nasally administered ketamine provides rapid and effective pain relief. Ketamine was well tolerated in these studies, side effects were transient and did not require treatment. 36,37 Results are promising, but nasal administration has its difficulties too. Intranasal administration irritates nasal mucosa and causes discomfort. Excessive mucus production, nose bleeds or destruction of nasal mucosa reduce effectiveness of a drug given intranasally. Administration in nebulized, inhaled form could provide without these problems but with same advantages as in intranasal administration.

Early on, ketamine has been observed to possess bronchodilatory effects. 32 Ketamine increases pulmonary compliance, decreases airway resistance and bronchospasm most likely by increasing catecholamine release, thus raising ß2-adrenergic stimulation and additionally by inhibiting vagal stimulation. 32,33

Inhaled nebulised ketamine has been investigated in an experimental animal model for the treatment of allergen-induced airway hyperresponsiveness and inflammation. 34 In that study alveolar ketamine was observed to suppress allergen-mediated airway hyperreactivity and airway inflammation. In another experimental study, the application of S(+)-ketamine in fluid-instilled lungs of anesthetized rats reduced alveolar fluid clearance by decreasing amiloride-sensitive transepithelial Na+ -transport. 35

Currently, there are no human studies on the use of ketamine as an analgesic in the nebulised, inhaled form.

Objectives

The primary purpose of this study is to evaluate whether nebulised S(+)-ketamine carries potential as a an analgesic bypassing first pass metabolism and without the need for intravenous access. Secondary aim is to assess the duration of analgesia obtained by nebulized S-ketamine. Thirdly, the aim is to evaluate whether inhaled nebulized ketamine decreases the need for rescue analgesia during PACU care.

Our hypothesis is that inhaled ketamine provides pain relief, which will be observed as lower numerical rating scale (NRS) values after ketamine administration.

Material and methods

Subjects

The subjects are recruited among patients coming in for a surgical intervention (orthopedic, gastrointestinal, plastic or urologic surgery) and needing further observation in postoperative care unit (PACU).

It was calculated that sample size of 8 subjects per group would be required to achieve statistical power of 80% and detect a difference of 3 units in NRS-values with standard deviation of 2 units and type I error of 5%. To prepare for possible dropouts, total of 20 subjects will be recruited (10 in each group).

Inclusion criteria

* male
* 18-65 years
* PACU care after general anaesthesia

Exclusion criteria

* female
* asthma
* chronic obstructive pulmonary disease
* diabetes mellitus
* unstable angina pectoris
* high intracranial pressure
* elevated intraocular pressure
* neurosurgery
* epidural or spinal analgesia
* history of long term pain state
* poor co-operation

Research methods

The study will be conducted as a double blind placebo-controlled crossover trial. A crossover design is chosen in order to reduce the incidence of confounding factors.

When the patients arrive at the PACU, monitoring will be commenced. Non-invasive blood pressure (NIBP), blood oxygen saturation (SpO2), 3-lead electrocardiogram (EKG), respiratory rate and Glasgow Coma Scale (GCS) will be monitored and recorded at 3 minute intervals throughout the protocol, otherwise every 15 minutes. The subjects will be observed for changes in neuropsychological status including behavior, sensory perception and pupillary status. Also respiratory patterns and salivation will be observed. Peak expiratory flow (PEF) will be measured before and within 5 minutes after exposure to study drugs.

Patients will receive either nebulized placebo (i.e. saline) or ketamine (Ketanest-S) when they require pain alleviation in the PACU. Dosage of ketamine is 1 mg/kg 36. Patients will be randomized into two groups so that other group's first inhalation contains ketamine and second inhalation placebo and in the opposite order. Neither the subjects nor the researchers know in which order preparations are administered. A person not involved in the study will prepare drugs beforehand and label them with A or B. Order of preparations will be determined using sequentially numbered, sealed opaque envelopes containing order in which preparations are given (either A B or B A). Envelope will be opened once patient arrives to PACU.

Inhalations will be given sequentially when the patient asks for pain medication. Subjects will receive two inhalations in total. Time between the inhalations will be measured in order to find out whether the analgesia after S-ketamine lasts for a longer time period than after placebo. The second inhalation serves as the rescue medication after the first inhalation, and may be dosed after three minutes after the first inhalation if not a significant reduction of pain is achieved in the NRS scale (>3 points). After the second inhalation, the pain of the patient is treated according to the clinical needs and following the protocol designed by the anaesthesiologist responsible for the patient. In our hospital iv oxycodone 1-4mg is used if suitable.

Before and after each drug administration the intensity of pain will be rated using a numerical rating scale (NRS) of 0 to 10 (0 = no pain, 10 = worst imaginable pain). Besides evaluating spontaneous postoperative pain, pain will be induced with pinprick test. Pinprick test is performed by sticking subject's arm with a sharp wooden toothpick. After drug administration, pricking will be carried on continuously rating pain intensity, until NRS-values are in the same level as in baseline. Time from start to the time when baseline NRS-value is reached, will be measured to estimate duration of analgesia.

Adverse effects will be evaluated using Side Effects Rating Scale for Dissociative Anesthetics (SERSDA). Patients will be contacted 24 hours after completing the study and queried about possible adverse effects and their severity using SERSDA. Side effects include fatigue, dizziness, nausea, headache, feeling of unreality, changes in hearing and vision, mood change, generalized discomfort and hallucination. Severity of side effects is rated on scale of 0 to 4 (0 = no change, 4 = very bothersome).

Data analysis

SPSS-program will be used for statistical analysis. Non-parametric tests will be applied in the analysis. P-values < 0,05 will be considered as statistically significant.

Ethical considerations

Guidelines of Good Clinical Practice will be followed 38. The study is conducted in volunteers in a controlled PACU setting. A written, informed consent is required for participation. Withdrawal from the study protocol is allowed at any point with intention to treat analysis applied and it will not affect the patient's treatment at the hospital. The study will be monitored.

Participants will not be harmed in the study. The minimal intensity of painful stimuli necessary for obtaining the study goals will be used and are performed routinely: the NIBP during the surgery every five minutes and in the PACU every 15 minutes, the pinprick when evaluating the level of postoperative analgetic treatment. Potential risks will be minimized by closely monitoring the subjects for the whole duration of the study. PACU personnel is prepared in case of any adverse effects occur.

All data gathered in this study will be treated with confidentiality and analyzed on a group level. An identification number (ID) will be given and the names of participants will be removed to ensure anonymity. Only members of the research group will have access to participants' identity information. All data will be stored in a locked, fireproof cabinet. Only researchers will have access to the data and the study code.

Implementation

Timetable

Recruiting the study subjects will start as soon as ethical and National Agency of Medicines (FIMEA) processes are completed, aim at early fall 2014. All data will be collected and analyzed by 2017.

Budget

Funding will be applied from FinnHEMS (Finnish Helicopter Emergency Medicine Service).

Distribution of work

Results of this study will be published in an international journal and as a part of doctoral thesis of Suvi-Maria Seppänen.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18-65 years of age
* PACU care after general anesthesia

Exclusion Criteria:

* female
* asthma
* COPD
* diabetes mellitus
* unstable angina pectoris
* high intracranial pressure
* elevated intraocular pressure
* neurosurgery
* epidural or spinal analgesia
* history of long-term pain state
* poor co-operation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Potential of S(+)-ketamine as an analgesic in the nebulised form | 3 minutes
  TIme measured for the second request of analgesia. 3 minutes is the anticipated duration of analgesia achieved by nebulised s-ketamine.

SECONDARY OUTCOMES:
Duration of analgesia | 10 minutes
  Duration of analgesia will be assessed by pin prick and will be measured in minutes and stopped when the NRS to pin prick equals base level measurement.
Duration of need for PACU care | 3 hours
  When the patient is qualified for returning to the ward, the time is marked.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Kämäräinen, MD, PhD, Principal Investigator — Pirkanmaa District Hospital, Department of Emergency Medicine
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clements JA, Nimmo WS. Pharmacokinetics and analgesic effect of ketamine in man. Br J Anaesth. 1981 Jan;53(1):27-30. doi: 10.1093/bja/53.1.27. PMID 7459184
- [Background] DOMINO EF, CHODOFF P, CORSSEN G. PHARMACOLOGIC EFFECTS OF CI-581, A NEW DISSOCIATIVE ANESTHETIC, IN MAN. Clin Pharmacol Ther. 1965 May-Jun;6:279-91. doi: 10.1002/cpt196563279. No abstract available. PMID 14296024
- [Background] Craven R. Ketamine. Anaesthesia. 2007 Dec;62 Suppl 1:48-53. doi: 10.1111/j.1365-2044.2007.05298.x. PMID 17937714
- [Background] Aan Het Rot M, Zarate CA Jr, Charney DS, Mathew SJ. Ketamine for depression: where do we go from here? Biol Psychiatry. 2012 Oct 1;72(7):537-47. doi: 10.1016/j.biopsych.2012.05.003. Epub 2012 Jun 16. PMID 22705040
- [Background] Aroni F, Iacovidou N, Dontas I, Pourzitaki C, Xanthos T. Pharmacological aspects and potential new clinical applications of ketamine: reevaluation of an old drug. J Clin Pharmacol. 2009 Aug;49(8):957-64. doi: 10.1177/0091270009337941. Epub 2009 Jun 22. PMID 19546251
- [Background] Klepstad P, Maurset A, Moberg ER, Oye I. Evidence of a role for NMDA receptors in pain perception. Eur J Pharmacol. 1990 Oct 23;187(3):513-8. doi: 10.1016/0014-2999(90)90379-k. PMID 1963598
- [Background] Arendt-Nielsen L, Nielsen J, Petersen-Felix S, Schnider TW, Zbinden AM. Effect of racemic mixture and the (S+)-isomer of ketamine on temporal and spatial summation of pain. Br J Anaesth. 1996 Nov;77(5):625-31. doi: 10.1093/bja/77.5.625. PMID 8957979
- [Background] Dal D, Celebi N, Elvan EG, Celiker V, Aypar U. The efficacy of intravenous or peritonsillar infiltration of ketamine for postoperative pain relief in children following adenotonsillectomy. Paediatr Anaesth. 2007 Mar;17(3):263-9. doi: 10.1111/j.1460-9592.2006.02095.x. PMID 17263742
- [Background] Chong C, Schug SA, Page-Sharp M, Jenkins B, Ilett KF. Development of a sublingual/oral formulation of ketamine for use in neuropathic pain: Preliminary findings from a three-way randomized, crossover study. Clin Drug Investig. 2009;29(5):317-24. doi: 10.2165/00044011-200929050-00004. PMID 19366273
- [Background] Christensen K, Rogers E, Green GA, et al. Safety and efficacy of intranasal ketamine for acute postoperative pain. Acute Pain. 2007;9(4):183-192.
- [Background] Zhu MM, Zhou QH, Zhu MH, Rong HB, Xu YM, Qian YN, Fu CZ. Effects of nebulized ketamine on allergen-induced airway hyperresponsiveness and inflammation in actively sensitized Brown-Norway rats. J Inflamm (Lond). 2007 May 4;4:10. doi: 10.1186/1476-9255-4-10. PMID 17480224
- [Background] Johansson J, Sjoberg J, Nordgren M, Sandstrom E, Sjoberg F, Zetterstrom H. Prehospital analgesia using nasal administration of S-ketamine--a case series. Scand J Trauma Resusc Emerg Med. 2013 May 14;21:38. doi: 10.1186/1757-7241-21-38. PMID 23672762
- [Background] European Medicines Agency. Guideline for good clinical practice 2002. www.ema.com.eu. Accessed 8/1, 2012.